CLINICAL TRIAL: NCT03380624
Title: Tear Lipid Layer Thickness With Emollient Eye Drops
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Jennifer Fogt, Associate Clinical Professor - Practice, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2016H0354
Record Dates: First submitted 2017-04-05; First posted 2017-12-21 (Actual); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Double masked, randomized
Who Masked: Participant, Outcomes Assessor
Masking Description: Investigator instills eye drop masked to participant. While this is a single arm study in that all participants receive both eye drops, the order in which they are used is randomized and masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Refresh Optive, then Refresh Optive MEGA-3 (Experimental): Participants first utilized one drop of Refresh Optive in each eye before taking lipid layer thickness measurements occurring at 15 minutes and 1 hour after instillation. After a washout period, they returned to repeat the testing using one drop of Refresh Optive MEGA-3 before taking lipid layer thickness measurements.
  .
  Interventions: Drug: Refresh Optive; Drug: Refresh Optive MEGA-3
- Refresh Optive MEGA-3, then Refresh Optive (Experimental): Participants first utilized one drop of Refresh Optive MEGA-3 in each eye before taking lipid layer thickness measurements occurring at 15 minutes and 1 hour after instillation. After a washout period, they returned to repeat the testing using one drop of Refresh Optive before taking lipid layer thickness measurements.
  Interventions: Drug: Refresh Optive; Drug: Refresh Optive MEGA-3

INTERVENTIONS:
Drug: Refresh Optive — Lubricate and hydrating relief of eye dryness investigational lubricant eye drop is based on carboxymethylcellulose
Drug: Refresh Optive MEGA-3 — Lubricate and hydrating relief of eye dryness investigational lubricant eye drop is based on carboxymethylcellulose and with flaxseed oil and trehalose

SUMMARY:
Crossover comparison of lipid layer thickness with two artificial tear formulations

DETAILED DESCRIPTION:
This study will objectively evaluate two US Monograph lubricant eyedrop formulations (Allergan, plc). Refresh Optive ADVANCED will be compared to an investigational formula with additional compendial ingredients (Refresh Optive MEGA 3) in subjects with dry eye symptoms and lipid layer thickness < 75 nm at baseline in a randomized, cross-over (masked subject) design. We seek to objectively evaluate the increase in lipid layer thickness from baseline at 15 minutes and 1 hour after each eye drop has been instilled. The Stroboscopic Video Color Microscope of King-Smith is used for non-invasive lipid layer thickness measurement.

ELIGIBILITY:
Inclusion Criteria:

* Age - at least 30 years

  * Good general health (defined by medication use that has not changed within the last month and the absence of medical conditions or treatments that are deemed confounding to the data as determined by the PI)
  * Ability to give informed consent
  * Willing to spend time for the study; approximately one hour for a screening visit and additional 4 hours for the study assessments. Study assessment will be conducted over 2 visit days, approximately 1 1/2 hours per day.
  * Either gender
  * Any racial or ethnic origin
  * Stroboscopic Video Color Microscope tear lipid thickness ≤ 75 nm

Exclusion Criteria:

* Use of any ocular prescription medication (such as but not limited to, glaucoma medications, anti-inflammatory eye drops and Restasis) used within 14 days of the screening visit or started prior to the measurement visit(s).

  * Currently having punctal plugs inserted in lacrimal puncta
  * Current eye disease, infection or inflammation that affects the surface of the eye such as, but not limited to moderate or greater blepharitis and ocular allergy. Clinically significant (active treatment) of blepharitis, Sjogren's disease or other systemic disease that could influence Meibomian Gland Dysfunction, corneal, conjunctival, or eyelid abnormalities that could influence lipid layer thickness, conjunctivitis of any cause, ocular infection or systemic medication such as diuretics or drugs that could influence tear secretion, or sensitivity to any of the ingredient in the eye drop being tested,
  * Past eye surgery, such as, but not limited to, refractive surgery. Subjects who have had cataract removal surgery more than one year ago, but less than 10 years ago may be considered as potential subjects.
  * Female subjects may not be pregnant or lactating. (Subject will be asked to self report these conditions.)
  * Infectious diseases (for example, hepatitis, tuberculosis) or an immuno-suppressive disease (for example, HIV). (Subjects will be asked to self-report these conditions.)
  * Inability to complete the screening and examination
  * Inability to provide analyzable data. For example, subjects who cannot keep their eye open during the entire measurement interval (due to early blinking) or provide a readable eye image (due to eyelid laxity) or cannot sit still for 1 minute.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Fogt, OD MS, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants were found to be ineligible after completing the baseline visit.
Groups:
- Refresh Optive Then Refresh Optive MEGA 3; Refresh Optive MEGA 3 Then Refresh Optive: The subjects are randomly assigned to one drop of Refresh Optive or Refresh Optive MEGA followed by measurement of lipid layer thickness at 15 minutes and 1 hour After which there is a washout period before Visit 2 - in which the measurements were repeated with the other eye drop.
Period: Overall Study
Arm/Group | Refresh Optive Then Refresh Optive MEGA 3 | Refresh Optive MEGA 3 Then Refresh Optive
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 21 subjects were enrolled. 19 completed both arms. At baseline, tear lipid layer thickness was assessed. Anyone with a tear lipid layer thickness greater than 75 nm were ineligible.
Groups:
- Refresh Optive and Refresh Optive MEGA: The subjects are randomly assigned to Refresh Optive or Refresh Optive MEGA (Omega 3) with measurements of lipid layer thickness following at 15 minutes and 1 hour.
  After which there is a washout period before proceeding to the second eye drop at visit 2.
  Refresh Optive: Lubricate and hydrating relief of eye dryness investigational lubricant eye drop is based on carboxymethylcellulose
  Refresh Optimum OMEGA 3: Lubricate and hydrating relief of eye dryness investigational lubricant eye drop is based on carboxymethylcellulose and with flaxseed oil and trehalose
  *All subjects completed both arms in this crossover study
Arm/Group | Refresh Optive and Refresh Optive MEGA
Number analyzed (Participants) | 19
Age, Customized [Count of Participants; unit: Participants]
  Age 30 to 65 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Lipid layer thickness [Mean (Standard Deviation); unit: nm] | 40.9 (10.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Tear Lipid Layer Thickness
Description: Change in tear lipid layer thickness
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: nm
Groups:
- Refresh Optive: Participants were first randomized to have 1 drop of Refresh Optive instilled in each eye with measurements of lipid layer thickness following at 15 minutes and 1 hour.
  After which there is a washout period before proceeding to a second visit in which Refresh Optive MEGA-3 was utilized and the measurements were repeated.
  Refresh Optive: Lubricate and hydrating relief of eye dryness investigational lubricant eye drop is based on carboxymethylcellulose
  Refresh Optimum OMEGA 3: Lubricate and hydrating relief of eye dryness investigational lubricant eye drop is based on carboxymethylcellulose and with flaxseed oil and trehalose
  *All subjects completed both arms in this crossover study
- Refresh Optive MEGA-3: Participants were first randomized to have 1 drop of Refresh Optive MEGA-3 instilled in each eye with measurements of lipid layer thickness following at 15 minutes and 1 hour.
  After which there is a washout period before proceeding to a second visit in which Refresh Optive was utilized and the measurements were repeated.
Arm/Group | Refresh Optive | Refresh Optive MEGA-3
Number analyzed (Participants) | 19 | 19
nm | 4.8 (14.9) | 8.8 (11.5)

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- Refresh Optive; Refresh Optive MEGA: The subjects are randomly assigned to Refresh Optive or Refresh Optive MEGA (Omega 3) with measurements of lipid layer thickness following at 15 minutes and 1 hour.
  After which there is a washout period before proceeding to the second eye drop at visit 2.
  Refresh Optive: Lubricate and hydrating relief of eye dryness investigational lubricant eye drop is based on carboxymethylcellulose
  Refresh Optimum OMEGA 3: Lubricate and hydrating relief of eye dryness investigational lubricant eye drop is based on carboxymethylcellulose and with flaxseed oil and trehalose
  *All subjects completed both arms in this crossover study
Arm/Group | Refresh Optive | Refresh Optive MEGA
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT03380624/Prot_000.pdf